CLINICAL TRIAL: NCT06773234
Title: Evaluation of the Dental Educational Environment in Upper Egypt Using the DREEM Tool: a Cross-Sectional Study
Brief Title: Evaluation of the Dental Educational Environment Using the DREEM Tool
Status: Recruiting | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Shereen Shaaban, Lecturer of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Beni-Suef University., Beni-Suef University
Other Study IDs: # REC-FDBSU/05122024-02/MS
Record Dates: First submitted 2024-12-31; First posted 2025-01-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Educational Problems
Keywords: Educational Environment; DREEM Tool
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- students from Faculty of Dentistry, Beni-Suef University: students from different educational levels in the Faculty of Dentistry, Beni-Suef University
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — DREEM Tool

SUMMARY:
This Cross-Sectional Study aims to evaluate the dental educational environment in Upper Egypt using the Dundee Ready Education Environment Measure (DREEM) Questionnaire.

DETAILED DESCRIPTION:
This Cross-Sectional Study aims to evaluate the dental educational environment in Upper Egypt using the Dundee Ready Education Environment Measure (DREEM) Questionnaire. The questionnaire will be sent to students in Faculty of Dentistry, Beni-Suef University to assess their perception of the educational environment.

ELIGIBILITY:
Inclusion Criteria:

* Students registered in the Faculty of Dentistry, Beni-Suef University

Exclusion Criteria:

- Students registered in any dental school other than the Faculty of Dentistry, Beni-Suef University.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: students registered in the Faculty of Dentistry, Beni-Suef University
Sampling Method: Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of dental students' perception of the educational environment. | 3 months
  Outcome Measuring Unit is 5 Likert scale scores as follows Strongly agree 4, Agree 3, Unsure 2, Disagree 1, and Strongly disagree 0

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Mustafa, Principal Investigator — Lecturer of Pediatric Dentistry and Dental Public Health Faculty of Dentistry, Beni-Suef University.
Locations (1):
- Faculty of Dentistry, Beni-Suef University., Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No